CLINICAL TRIAL: NCT00375583
Title: Effect of Albendazole Dose and Interval on Wuchereria Bancrofti Microfilarial Clearance in India: A Randomized, Open Label Study
Brief Title: Effect of Albendazole Dose on Clearance of Filarial Worms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Tuberculosis Research Centre, India (Other Government)
Responsible Party: Thomas B. Nutman, M.D./National Institute of Allergy and Infectious Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999906244; 06-I-N244
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-28

CONDITIONS: Lymphatic Filariasis; Wuchereria Bancrofti Infection
Keywords: Lymphatic Filariasis; Diethylcarbamazine; Microfilariae; Helminths; Nematode
MeSH Terms: conditions — Elephantiasis, Filarial; Enterobiasis

INTERVENTIONS:
Drug: DEC/Albendazole

SUMMARY:
This study, conducted in Chennai, India, will determine whether a new treatment regimen of albendazole and diethylcarbamazine for lymphatic filariasis can eliminate the disease more quickly than the standard regimen. Lymphatic filariasis is caused by infection with very small filarial worms, particulalry Wuchereria bancroti, that are spread by mosquitoes. The infection can lead to swelling of the arms, legs, breast and scrotum and can progress to permanent swelling of the legs or arms called elephantiasis. The study will see if a higher and more frequent dose of albendazole is better at clearing filarial worms from the blood than the current treatment.

Healthy people between 18 and 55 years of age who are in good health and who are infected with Wuchereria bancrofti may be eligible for this 28-month study. Candidates must be willing to spend 4 days in the Government General Hospital in Chennai, India, at the beginning of the study. They are screened with a medical history, a brief physical examination, ultrasound (picture generated by sound waves) of the groin or chest, and blood tests to check for infection with Wuchereria bancrofti and to measure white blood cell counts.

Participants undergo the following procedures:

-4-day hospitalization

Random assignment to receive either standard treatment (400 mg albendazole and 300 mg DEC given once a year for 2 years) or the experimental regimen (800 mg albendazole and 300 mg DEC given twice a year for 2 years)

Urine pregnancy test for women of childbearing age

Receive first treatment dose

Monitoring for symptoms

-6-month outpatient visit

Short history, physical examination and blood test

Second treatment dose for subjects receiving 800 mg albendazole

Urine pregnancy test for women of childbearing age

-1-year outpatient visit

Short history, physical examination and blood test

Second or third treatment dose, depending on treatment group

Repeat ultrasound in subjects whose first ultrasound detected adult worm

Urine pregnancy test for women of childbearing age

-18-month outpatient visit

Short history, physical examination and blood test

Fourth treatment dose for subjects receiving 800 mg albendazole

Urine pregnancy test for women of childbearing age

-24-month outpatient visit

Short history, physical examination and blood test

Final dose of albendazole and DEC at standard doses

Repeat ultrasound in subjects whose first ultrasound detected adult worms

Urine pregnancy test for women of childbearing age

DETAILED DESCRIPTION:
Albendazole and diethylcarbamazine (DEC) are currently used in combination for annual mass treatment of lymphatic filariasis in all parts of the world except Africa. Although the drugs have been donated, the cost of such programs is very high and has proven to be a major impediment to the success of programs in many countries with limited financial resources. Data from albendazole treatment of other filarial infections and one study comparing single to multi-dose DEC/albendazole in lymphatic filariasis suggest that increased dose and/or frequency of albendazole dosing may be more effective in clearing microfilariae. In this study, 50 volunteers with microfilaremic Wuchereria bancrofti infection will be randomized to receive standard annual therapy (albendazole 400 mg + DEC 300 mg) or semiannual therapy with an increased albendazole dose (albendazole 800 mg + DEC 300 mg). Microfilarial levels, as well as measures of adult worm burden (circulating antigen, ultrasound identification of adult worm nests) will be followed every six months for two years to determine whether the higher dose, more frequent regimen is more effective.

ELIGIBILITY:
* INCLUSION CRITERIA (SCREENING):

Age 18 years to 55 years inclusive.

Both genders.

Not pregnant or breastfeeding by history.

If selected, subject must be willing to spend 3 days on the Clinical Trials Unit of the Government General Hospital, Chennai India.

If selected, subject must be willing to undergo nighttime blood draws every 6 months for 2 years.

If selected, agree to have blood stored for future studies.

Ability to understand and sign the informed consent.

EXCLUSION CRITERIA (SCREENING):

Non-volunteers.

Age less than 18 years or greater than 55 years.

Pregnant or breastfeeding by history.

INCLUSION (TREATMENT):

Age 18 years to 55 years.

Men and non-pregnant or non-breastfeeding women.

Microfilarial levels greater than 50 mf/ml.

Willingness to spend 3 days on the Clinical Trials Unit of the Government General Hospital, Chennai India.

Willingness to undergo nighttime blood draws every 6 months for 2 years.

Ability to understand and sign the informed consent.

Hb levels for inclusion greater than 9 g/dL.

Normal Cr, ALT.

Willingness to have blood stored for future studies.

EXCLUSION (TREATMENT):

Non-volunteers.

Age less than 18 years or greater than 55 years.

Pregnancy or breast-feeding.

Hgb less than or equal to 9 g/dL.

Cr greater than 1.2/100 ml.

ALT greater than 30 U.

Alcohol consumption of more than 2 beers or other alcohol-containing drink/day within a week of each drug administration.

Temperature greater than 37.5 degrees C.

Serious medical illness.

History of benzimidazole allergy.

History of DEC allergy.

Use of albendazole or DEC within past 6 months.

Unwillingness to comply with required study visits.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-09-09; Primary Completion 2011-04-28 (Actual); Study Completion 2011-04-28 (Actual)

PRIMARY OUTCOMES:
Microfilarial levels. | 12 months.

SECONDARY OUTCOMES:
Adult worm burden. | 12 and 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuberculosis Research Centre, Chennai, India

REFERENCES:
- [Background] Adjepon-Yamoah KK, Edwards G, Breckenridge AM, Orme ML, Ward SA. The effect of renal disease on the pharmacokinetics of diethylcarbamazine in man. Br J Clin Pharmacol. 1982 Jun;13(6):829-34. doi: 10.1111/j.1365-2125.1982.tb01874.x. PMID 7093114
- [Background] Andrade LD, Medeiros Z, Pires ML, Pimentel A, Rocha A, Figueredo-Silva J, Coutinho A, Dreyer G. Comparative efficacy of three different diethylcarbamazine regimens in lymphatic filariasis. Trans R Soc Trop Med Hyg. 1995 May-Jun;89(3):319-21. doi: 10.1016/0035-9203(95)90561-8. PMID 7660449
- [Background] Amaral F, Dreyer G, Figueredo-Silva J, Noroes J, Cavalcanti A, Samico SC, Santos A, Coutinho A. Live adult worms detected by ultrasonography in human Bancroftian filariasis. Am J Trop Med Hyg. 1994 Jun;50(6):753-7. doi: 10.4269/ajtmh.1994.50.753. PMID 8024070